CLINICAL TRIAL: NCT03025763
Title: Craniosynostosis Network
Brief Title: Network Of Clinical Research Studies On Craniosynostosis, Skull Malformations With Premature Fusion Of Skull Bones
Status: Active, not recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Ethylin Wang Jabs, Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 13-0147; P01HD078233 (NIH)
Record Dates: First submitted 2017-01-17; First posted 2017-01-20 (Estimated); Last update posted 2025-01-02 (Actual); Status verified 2024-12

CONDITIONS: Craniosynostosis
Keywords: Craniosynostosis; Bone; Birth Defect; Congenital Anomaly; Malformation; Genetics; Genomics; Skull; Human; Mouse; Imaging; Cell Biology; Induced Pluripotent Stem Cells; System Biology
MeSH Terms: conditions — Craniosynostoses; Congenital Abnormalities | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Saliva, blood, white blood cells, DNA, RNA, and generated induced pluripotent stem cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Coronal Nonsyndromic Craniosynostosis, trios: Participants with diagnosis of coronal, nonsyndromic craniosynostosis including affected and unaffected biological parents
  Interventions: Other: Craniosynostosis Network Environmental Survey; Other: 2D/3D Photography; Procedure: Buccal Swab Cell Sampling; Procedure: Blood sampling; Procedure: Skin Biopsy; Procedure: Tissues from a Clinically Indicated Procedure; Procedure: Pre-operative CT Scan Image Files.
- Coronal, nonsyndromic craniosynostosis: Participants with coronal, nonsyndromic craniosynostosis when biological parents are not available
  Interventions: Other: Craniosynostosis Network Environmental Survey; Other: 2D/3D Photography; Procedure: Buccal Swab Cell Sampling; Procedure: Blood sampling; Procedure: Skin Biopsy; Procedure: Tissues from a Clinically Indicated Procedure; Procedure: Pre-operative CT Scan Image Files.
- Unaffected controls: Unaffected controls who may have undergone clinically indicated craniofacial surgery for trauma or conditions other than craniosynostosis or bone disease
  Interventions: Other: Craniosynostosis Network Environmental Survey; Other: 2D/3D Photography; Procedure: Buccal Swab Cell Sampling; Procedure: Blood sampling; Procedure: Skin Biopsy; Procedure: Tissues from a Clinically Indicated Procedure; Procedure: Pre-operative CT Scan Image Files.

INTERVENTIONS:
Other: Craniosynostosis Network Environmental Survey — Questionnaire is administered to the mothers of affected participants regarding medical history and environmental exposures during pregnancy, delivery, and neonatal period. Optional.
Other: 2D/3D Photography — Full frontal and lateral face and other parts of the body may be taken for dysmorphic assessment. There is the risk of identification and loss of confidentiality. Optional.
Procedure: Buccal Swab Cell Sampling — One or more swabs, like a Q-tip (for children), or saliva collection kit (for adults) will be used to collect buccal cells. With a swab, they will brush the inside of the mouth several times. With saliva collection kit, they will collect their saliva by spitting into a container several times using a commercially available saliva collection kit. Required.
Procedure: Blood sampling — Venipuncture so that one teaspoon to tablespoons (1-20 ml.) of blood is collected. The volume drawn will be dependent on the age and size of the child. Minimal amounts may be required for DNA, but to establish a lymphoblastoid or iPS cell line at least 3 to 10 ml will be required independent of age. In the case of an infant, if 3 to 10 ml cannot be obtained, then a lymphoblastoid or iPS cell line will not be created. Optional.
Procedure: Skin Biopsy — For those who do not undergo surgery or the skin removal is not considered part of the surgical procedure. After proper cleaning, a piece of skin the size of a pencil eraser (about 4 mm or 1/8 inch in diameter) will be removed (using a circular blade or scalpel) from the arm (inside of arm or forearm in a spot that is as unnoticeable as possible). This area will be covered with a Band-Aid. No stitches are usually required. A crust will form and eventually fall off. Optional.
Procedure: Tissues from a Clinically Indicated Procedure — In some instances when there is discarded tissues and specimens (including skin and bone at the time of reconstructive craniofacial surgery), they will be collected by making arrangements with their physicians. Some of these tissues will be used to generate cell lines. Optional.
Procedure: Pre-operative CT Scan Image Files. — Optional for those who had a previous CT scan for a prior traumatic event.

SUMMARY:
Craniosynostosis (CS) is a common malformation occurring in ~4 per 10,000 live births in which the sutures between skull bones close too early, causing long-term problems with brain and skull growth. Infants with CS typically require extensive surgical treatment and may experience many perioperative complications, including hemorrhage and re-synostosis. Even with successful surgery, children can experience developmental and learning disabilities or vision problems. Most often, CS appears as isolated nonsyndromic CS (NSC). Of the several subtypes of CS, unilateral or bilateral fusion of the coronal suture is the second most common form of CS accounting for 20-30% of all NSC cases. The etiology of coronal NSC (cNSC) is not well understood, although the published literature suggests that it is a multifactorial condition. About 5-14% of coronal craniosynostosis patients have a positive family history, with a specific genetic etiology identified in >25% of cNSC cases, suggesting a strong genetic component in the pathogenesis of this birth defect. The causes for cNSC and its phenotypic heterogeneity remain largely unknown. An international team of investigators will generate large genomic and gene expression datasets on samples from patients with cNSC. State-of-the-art imaging, genetic, and developmental and systems biology approaches will be used to quantitatively model novel pathways and networks involved in the development of cNSC. Novel variant-, gene- and network-level analyses will be performed on the genomic data obtained from cNSC cases, their relatives, and controls to identify novel variants and genetic regions associated with cNCS. Quantitative, analytical, and functional validations of these predictions will provide insights into the etiology and possible therapeutic targets for CS and potentially other bone-related disorders.

DETAILED DESCRIPTION:
The long-term goal of the Program Project, Craniosynostosis Network, is to elucidate normal and abnormal craniofacial biology to ultimately improve the treatment of craniofacial disorders. Craniosynostosis and other skull abnormalities are among the most common human malformations usually requiring surgical and medical intervention. The Network will integrate three projects and two cores. Scientists with diverse expertise including anthropology, morphometry, imaging, birth defects, developmental biology, genetics, genomics, epidemiology, statistics, and systems biology will explore the determinants of the fate of the relevant mesenchymal progenitor cells, abnormalities in osteogenesis that contribute to global skull growth abnormality and premature closure of cranial sutures, especially the coronal suture. High quality genomic data will be obtained from patients with coronal nonsyndromic craniosynostosis (cNSC) and their available parents. Novel genome-wide variant-, gene- and network-level analyses will be performed on these families to identify novel variants and genetic regions associated with coronal craniosynostosis.

This study is a multi-center, open-enrollment, retrospective study, employing both family-based and case-control study designs.

Approximately 4000 cNSC patients, their family members, and controls will be recruited by Icahn School of Medicine at Mount Sinai and the majority will be recruited from the more than 10 collaborating institutions worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Cases with diagnosis of coronal
* Unaffected relatives of cases
* Unaffected controls including those who may have undergone clinically indicated craniofacial surgery for trauma or conditions other than craniosynostosis or bone disease. These individuals will be recruited at some of the other collaborating institutions, but not at Mount Sinai.

Individuals of any racial or ethnic group with the established or suspected clinical diagnosis of coronal, nonsyndromic craniosynostosis will be included in this study. Unaffected relatives, such as their biological parents and/or sibs, will also be included to contribute medical information and samples as negative controls for our study.

Exclusion Criteria:

* Those who fit the criteria, but who choose not to participate
* Those who do not meet the criteria.
* Other than children, no vulnerable individuals will be recruited, such as intellectual impaired individuals or prisoners.

Max Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with coronal nonsyndromic craniosynostosis (cNSC) and their relatives and controls (including noncraniosynostosis patients having neurosurgery for another surgical indication) will be included in this study. Approximately 4,000 individuals will participate of either gender and all ages, ethnicities, and race. All research subjects will be consented through approved IRB protocols at Icahn School of Medicine at Mount Sinai or respective collaborating institutions which will be governed by their own institutional IRB committees. Only de-identified medical information, CT scans, and samples from collaborating institutions will be shared with Mount Sinai.
Sampling Method: Non-Probability Sample
Enrollment: 2145 (Actual)
Dates: Start 2015-01-13 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Phenotype-genotype gene expression correlations | up to 5 years
  Phenotype-genotype-gene expression correlations among cohorts of cases of coronal nonsyndromic craniosynostosis and genotype-gene expression correlations among controls will be analyzed and compared.

SECONDARY OUTCOMES:
Incidence of gene mutations | up to 5 years
  gene mutations and variants may be found that are significantly associated with coronal nonsyndromic craniosynostosis

CONTACTS AND LOCATIONS:
Overall Officials: Ethylin Wang Jabs, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Inga Peter, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (20):
- United States (15):
  - The International Craniosynostosis Consortium at University of California at Davis, Davis, California
  - Yale University, Hartford, Connecticut
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - National Birth Defects Prevention Study at University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Birth Defect Registries of New York State, Albany, New York
  - New York University, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Pennsylvania State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Pennsylvania State University, University Park, Pennsylvania
  - Seton Family of Hospitals, Austin, Texas
  - Medical City Children's Hospital, Dallas, Texas
  - University of Texas at Southwestern, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
- France (2):
  - University of Bordeaux, Talence, Aquitaine
  - INSERM/ Hospital Necker-Enfants Malades, Paris, Cedex 14
- University Hospital Heidelberg, Heidelberg, Germany
- Hospital Sant Joan de Deu, Barcelona, Esplugues de Llobregat, Spain
- Oxford University, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Clinical results from chromosomal analysis and DNA mutation analysis performed in CLIA approved laboratories with standard clinical genetic counseling will be given to the patient upon request. Individual research results will be made available to the individual from the PI or their primary care physician (PCP) who has obtained preliminary results from the PI from our non-CLIA laboratory, as long as the PCP can confirm and validate the lab results through a CLIA approved lab before the results are given to the subjects.
Supporting Information: Study Protocol, ICF
Time Frame: Data with statistical analysis will become available with peer-reviewed publication
Access Criteria: Deidentified data will be deposited into public resource databases including whole genome sequencing data deposited in dbGAP with the identifier phs001806.v1.p1 and RNA-seq data deposited in Gene Expression Omnibus (GEO) with accession number GSE200492.

REFERENCES:
- [Background] Heuze Y, Holmes G, Peter I, Richtsmeier JT, Jabs EW. Closing the Gap: Genetic and Genomic Continuum from Syndromic to Nonsyndromic Craniosynostoses. Curr Genet Med Rep. 2014 Sep 1;2(3):135-145. doi: 10.1007/s40142-014-0042-x. PMID 26146596
- [Background] Heuze Y, Singh N, Basilico C, Jabs EW, Holmes G, Richtsmeier JT. Morphological comparison of the craniofacial phenotypes of mouse models expressing the Apert FGFR2 S252W mutation in neural crest- or mesoderm-derived tissues. Bone. 2014 Jun;63:101-9. doi: 10.1016/j.bone.2014.03.003. Epub 2014 Mar 13. PMID 24632501
- [Background] Heuze Y, Martinez-Abadias N, Stella JM, Arnaud E, Collet C, Garcia Fructuoso G, Alamar M, Lo LJ, Boyadjiev SA, Di Rocco F, Richtsmeier JT. Quantification of facial skeletal shape variation in fibroblast growth factor receptor-related craniosynostosis syndromes. Birth Defects Res A Clin Mol Teratol. 2014 Apr;100(4):250-9. doi: 10.1002/bdra.23228. Epub 2014 Feb 27. PMID 24578066
- [Background] Di Rocco F, Biosse Duplan M, Heuze Y, Kaci N, Komla-Ebri D, Munnich A, Mugniery E, Benoist-Lasselin C, Legeai-Mallet L. FGFR3 mutation causes abnormal membranous ossification in achondroplasia. Hum Mol Genet. 2014 Jun 1;23(11):2914-25. doi: 10.1093/hmg/ddu004. Epub 2014 Jan 12. PMID 24419316
- [Background] Justice CM, Yagnik G, Kim Y, Peter I, Jabs EW, Erazo M, Ye X, Ainehsazan E, Shi L, Cunningham ML, Kimonis V, Roscioli T, Wall SA, Wilkie AO, Stoler J, Richtsmeier JT, Heuze Y, Sanchez-Lara PA, Buckley MF, Druschel CM, Mills JL, Caggana M, Romitti PA, Kay DM, Senders C, Taub PJ, Klein OD, Boggan J, Zwienenberg-Lee M, Naydenov C, Kim J, Wilson AF, Boyadjiev SA. A genome-wide association study identifies susceptibility loci for nonsyndromic sagittal craniosynostosis near BMP2 and within BBS9. Nat Genet. 2012 Dec;44(12):1360-4. doi: 10.1038/ng.2463. Epub 2012 Nov 18. PMID 23160099
- [Background] Heuze Y, Martinez-Abadias N, Stella JM, Senders CW, Boyadjiev SA, Lo LJ, Richtsmeier JT. Unilateral and bilateral expression of a quantitative trait: asymmetry and symmetry in coronal craniosynostosis. J Exp Zool B Mol Dev Evol. 2012 Mar;318(2):109-22. doi: 10.1002/jezb.21449. PMID 22532473
- [Background] Martinez-Abadias N, Heuze Y, Wang Y, Jabs EW, Aldridge K, Richtsmeier JT. FGF/FGFR signaling coordinates skull development by modulating magnitude of morphological integration: evidence from Apert syndrome mouse models. PLoS One. 2011;6(10):e26425. doi: 10.1371/journal.pone.0026425. Epub 2011 Oct 28. PMID 22053191
- [Background] Heuze Y, Boyadjiev SA, Marsh JL, Kane AA, Cherkez E, Boggan JE, Richtsmeier JT. New insights into the relationship between suture closure and craniofacial dysmorphology in sagittal nonsyndromic craniosynostosis. J Anat. 2010 Aug;217(2):85-96. doi: 10.1111/j.1469-7580.2010.01258.x. Epub 2010 Jun 22. PMID 20572900
- [Background] Wang Y, Sun M, Uhlhorn VL, Zhou X, Peter I, Martinez-Abadias N, Hill CA, Percival CJ, Richtsmeier JT, Huso DL, Jabs EW. Activation of p38 MAPK pathway in the skull abnormalities of Apert syndrome Fgfr2(+P253R) mice. BMC Dev Biol. 2010 Feb 22;10:22. doi: 10.1186/1471-213X-10-22. PMID 20175913
- [Background] Percival CJ, Kawasaki K, Huang Y, Weiss KM, Jabs EW, Li R, Richtsmeier JT. Building Bones. Percival CJ, Richtsmeier JT, editors. Cambridge. Cambridge University Press; 2017. Chapter 2, The contribution of angiogenesis to variation in bone development and evolution; 26-51p.
- [Background] Kawasaki K, Richtsmeier JT. Building Bones. Percival CJ, Richtsmeier JT, editors. Cambridge. Cambridge University Press; 2017. Chapter 3, Association of the chondrocranium and dermatocranium in early skull development; 52-78p.
- [Background] Kawasaki K, Richtsmeier J. Building Bones. Percival CJ, Richtsmeier JT, editors. Cambridge. Cambridge University Press; 2017. Chapter Appendix, Appendix to Chapter 3 ; 303-315p.
- [Background] Singh N, Dutka T, Reeves RH, Richtsmeier JT. Chronic up-regulation of sonic hedgehog has little effect on postnatal craniofacial morphology of euploid and trisomic mice. Dev Dyn. 2016 Feb;245(2):114-22. doi: 10.1002/dvdy.24361. Epub 2015 Dec 6. PMID 26509735
- [Background] Trainor PA, Richtsmeier JT. Facing up to the challenges of advancing Craniofacial Research. Am J Med Genet A. 2015 Jul;167(7):1451-4. doi: 10.1002/ajmg.a.37065. Epub 2015 Mar 28. PMID 25820983
- [Background] Wilkie AOM, Johnson D, Wall SA. Clinical genetics of craniosynostosis. Curr Opin Pediatr. 2017 Dec;29(6):622-628. doi: 10.1097/MOP.0000000000000542. PMID 28914635
- [Background] Richtsmeier JT, Jones MC, Lozanoff S, Trainor PA. The Society for Craniofacial Genetics and Developmental Biology 37th annual meeting. Am J Med Genet A. 2015 Jul;167(7):1455-73. doi: 10.1002/ajmg.a.37012. Epub 2015 Mar 30. No abstract available. PMID 25820705
- [Background] Singh N, Dutka T, Devenney BM, Kawasaki K, Reeves RH, Richtsmeier JT. Acute upregulation of hedgehog signaling in mice causes differential effects on cranial morphology. Dis Model Mech. 2015 Mar;8(3):271-9. doi: 10.1242/dmm.017889. Epub 2014 Dec 24. PMID 25540129
- [Result] Flaherty K, Singh N, Richtsmeier JT. Understanding craniosynostosis as a growth disorder. Wiley Interdiscip Rev Dev Biol. 2016 Jul;5(4):429-59. doi: 10.1002/wdev.227. Epub 2016 Mar 22. PMID 27002187
- [Result] Ye X, Guilmatre A, Reva B, Peter I, Heuze Y, Richtsmeier JT, Fox DJ, Goedken RJ, Jabs EW, Romitti PA. Mutation Screening of Candidate Genes in Patients with Nonsyndromic Sagittal Craniosynostosis. Plast Reconstr Surg. 2016 Mar;137(3):952-961. doi: 10.1097/01.prs.0000479978.75545.ee. PMID 26910679
- [Result] Musy M, Flaherty K, Raspopovic J, Robert-Moreno A, Richtsmeier JT, Sharpe J. A quantitative method for staging mouse embryos based on limb morphometry. Development. 2018 Apr 5;145(7):dev154856. doi: 10.1242/dev.154856. PMID 29540505
- [Result] Heuze Y, Kawasaki K, Schwarz T, Schoenebeck JJ, Richtsmeier JT. Developmental and Evolutionary Significance of the Zygomatic Bone. Anat Rec (Hoboken). 2016 Dec;299(12):1616-1630. doi: 10.1002/ar.23449. PMID 27870340
- [Result] Motch Perrine SM, Stecko T, Neuberger T, Jabs EW, Ryan TM, Richtsmeier JT. Integration of Brain and Skull in Prenatal Mouse Models of Apert and Crouzon Syndromes. Front Hum Neurosci. 2017 Jul 25;11:369. doi: 10.3389/fnhum.2017.00369. eCollection 2017. PMID 28790902
- [Result] Lee C, Richtsmeier JT, Kraft RH. A COMPUTATIONAL ANALYSIS OF BONE FORMATION IN THE CRANIAL VAULT USING A COUPLED REACTION-DIFFUSION-STRAIN MODEL. J Mech Med Biol. 2017 Jun;17(4):1750073. doi: 10.1142/S0219519417500737. Epub 2017 May 29. PMID 29225392
- [Result] Lesciotto KM, Heuze Y, Jabs EW, Bernstein JM, Richtsmeier JT. Choanal Atresia and Craniosynostosis: Development and Disease. Plast Reconstr Surg. 2018 Jan;141(1):156-168. doi: 10.1097/PRS.0000000000003928. PMID 29280877
- [Result] Motch Perrine SM, Wu M, Stephens NB, Kriti D, van Bakel H, Jabs EW, Richtsmeier JT. Mandibular dysmorphology due to abnormal embryonic osteogenesis in FGFR2-related craniosynostosis mice. Dis Model Mech. 2019 May 30;12(5):dmm038513. doi: 10.1242/dmm.038513. PMID 31064775
- [Result] Norwood JN, Zhang Q, Card D, Craine A, Ryan TM, Drew PJ. Anatomical basis and physiological role of cerebrospinal fluid transport through the murine cribriform plate. Elife. 2019 May 7;8:e44278. doi: 10.7554/eLife.44278. PMID 31063132
- [Result] Lee C, Richtsmeier JT, Kraft RH. A coupled reaction-diffusion-strain model predicts cranial vault formation in development and disease. Biomech Model Mechanobiol. 2019 Aug;18(4):1197-1211. doi: 10.1007/s10237-019-01139-z. Epub 2019 Apr 20. PMID 31006064
- [Result] Sewda A, White SR, Erazo M, Hao K, Garcia-Fructuoso G, Fernandez-Rodriguez I, Heuze Y, Richtsmeier JT, Romitti PA, Reva B, Jabs EW, Peter I. Nonsyndromic craniosynostosis: novel coding variants. Pediatr Res. 2019 Mar;85(4):463-468. doi: 10.1038/s41390-019-0274-2. Epub 2019 Jan 14. PMID 30651579
- [Result] Lesciotto KM, Richtsmeier JT. Craniofacial skeletal response to encephalization: How do we know what we think we know? Am J Phys Anthropol. 2019 Jan;168 Suppl 67(Suppl 67):27-46. doi: 10.1002/ajpa.23766. PMID 30680710
- [Result] Flaherty K, Richtsmeier JT. It's about Time: Ossification Center Formation in C57BL/6 Mice from E12(-)E16. J Dev Biol. 2018 Dec 15;6(4):31. doi: 10.3390/jdb6040031. PMID 30558321
- [Result] Holmes G, O'Rourke C, Motch Perrine SM, Lu N, van Bakel H, Richtsmeier JT, Jabs EW. Midface and upper airway dysgenesis in FGFR2-related craniosynostosis involves multiple tissue-specific and cell cycle effects. Development. 2018 Oct 5;145(19):dev166488. doi: 10.1242/dev.166488. PMID 30228104
- [Result] Martinez-Abadias N, Mateu Estivill R, Sastre Tomas J, Motch Perrine S, Yoon M, Robert-Moreno A, Swoger J, Russo L, Kawasaki K, Richtsmeier J, Sharpe J. Quantification of gene expression patterns to reveal the origins of abnormal morphogenesis. Elife. 2018 Sep 20;7:e36405. doi: 10.7554/eLife.36405. PMID 30234486
- [Result] Holmes G, Zhang L, Rivera J, Murphy R, Assouline C, Sullivan L, Oppeneer T, Jabs EW. C-type natriuretic peptide analog treatment of craniosynostosis in a Crouzon syndrome mouse model. PLoS One. 2018 Jul 26;13(7):e0201492. doi: 10.1371/journal.pone.0201492. eCollection 2018. PMID 30048539
- [Result] Richtsmeier JT. A century of development. Am J Phys Anthropol. 2018 Apr;165(4):726-740. doi: 10.1002/ajpa.23379. No abstract available. PMID 29574839
- [Result] Starbuck JM, Cole TM 3rd, Reeves RH, Richtsmeier JT. The Influence of trisomy 21 on facial form and variability. Am J Med Genet A. 2017 Nov;173(11):2861-2872. doi: 10.1002/ajmg.a.38464. Epub 2017 Sep 21. PMID 28941128
- [Result] Weiss K, Buchanan A, Richtsmeier J. How are we made?: Even well-controlled experiments show the complexity of our traits. Evol Anthropol. 2015 Jul-Aug;24(4):130-6. doi: 10.1002/evan.21454. No abstract available. PMID 26267434
- [Result] Lee C, Richtsmeier JT, Kraft RH. A computational analysis of bone formation in the cranial vault in the mouse. Front Bioeng Biotechnol. 2015 Mar 19;3:24. doi: 10.3389/fbioe.2015.00024. eCollection 2015. PMID 25853124
- [Result] Pitirri MK, Richtsmeier JT, Kawasaki M, Coupe AP, Perrine SM, Kawasaki K. Come together over me: Cells that form the dermatocranium and chondrocranium in mice. Anat Rec (Hoboken). 2025 Jul;308(7):1972-1993. doi: 10.1002/ar.25295. Epub 2023 Jul 27. PMID 37497849
- [Result] Lesciotto KM, Tomlinson L, Leonard S, Richtsmeier JT. Embryonic and early postnatal cranial bone volume and tissue mineral density values for C57BL/6J laboratory mice. Dev Dyn. 2022 Jul;251(7):1196-1208. doi: 10.1002/dvdy.458. Epub 2022 Feb 7. PMID 35092111
- [Result] Pitirri MK, Durham EL, Romano NA, Santos JI, Coupe AP, Zheng H, Chen DZ, Kawasaki K, Jabs EW, Richtsmeier JT, Wu M, Motch Perrine SM. Meckel's Cartilage in Mandibular Development and Dysmorphogenesis. Front Genet. 2022 May 16;13:871927. doi: 10.3389/fgene.2022.871927. eCollection 2022. PMID 35651944
- [Result] Wu M, Kriti D, van Bakel H, Jabs EW, Holmes G. Laser Capture Microdissection of Mouse Embryonic Cartilage and Bone for Gene Expression Analysis. J Vis Exp. 2019 Dec 18;(154). doi: 10.3791/60503. PMID 31904019
- [Result] Kawasaki K, Mikami M, Goto M, Shindo J, Amano M, Ishiyama M. The Evolution of Unusually Small Amelogenin Genes in Cetaceans; Pseudogenization, X-Y Gene Conversion, and Feeding Strategy. J Mol Evol. 2020 Mar;88(2):122-135. doi: 10.1007/s00239-019-09917-0. Epub 2019 Nov 22. PMID 31754761
- [Result] Pitirri MK, Kawasaki K, Richtsmeier JT. It takes two: Building the vertebrate skull from chondrocranium and dermatocranium. Vertebr Zool. 2020 Apr;70(4):587-600. Epub 2020 Oct 28. PMID 33163116
- [Result] Holmes G, Gonzalez-Reiche AS, Lu N, Zhou X, Rivera J, Kriti D, Sebra R, Williams AA, Donovan MJ, Potter SS, Pinto D, Zhang B, van Bakel H, Jabs EW. Integrated Transcriptome and Network Analysis Reveals Spatiotemporal Dynamics of Calvarial Suturogenesis. Cell Rep. 2020 Jul 7;32(1):107871. doi: 10.1016/j.celrep.2020.107871. PMID 32640236
- [Result] Lam AS, Liu CC, Deutsch GH, Rivera J, Perkins JA, Holmes G, Jabs EW, Cunningham ML, Dahl JP. Genotype-Phenotype Correlation of Tracheal Cartilaginous Sleeves and Fgfr2 Mutations in Mice. Laryngoscope. 2021 Apr;131(4):E1349-E1356. doi: 10.1002/lary.29060. Epub 2020 Sep 4. PMID 32886384
- [Result] Singh R, Cohen ASA, Poulton C, Hjortshoj TD, Akahira-Azuma M, Mendiratta G, Khan WA, Azmanov DN, Woodward KJ, Kirchhoff M, Shi L, Edelmann L, Baynam G, Scott SA, Jabs EW. Deletion of ERF and CIC causes abnormal skull morphology and global developmental delay. Cold Spring Harb Mol Case Stud. 2021 Jun 11;7(3):a005991. doi: 10.1101/mcs.a005991. Print 2021 Jun. PMID 34117072
- [Result] Holmes G, Gonzalez-Reiche AS, Saturne M, Motch Perrine SM, Zhou X, Borges AC, Shewale B, Richtsmeier JT, Zhang B, van Bakel H, Jabs EW. Single-cell analysis identifies a key role for Hhip in murine coronal suture development. Nat Commun. 2021 Dec 8;12(1):7132. doi: 10.1038/s41467-021-27402-5. PMID 34880220
- [Result] Nicoletti P, Zafer S, Matok L, Irron I, Patrick M, Haklai R, Evangelista JE, Marino GB, Ma'ayan A, Sewda A, Holmes G, Britton SR, Lee WJ, Wu M, Ru Y, Arnaud E, Botto L, Brody LC, Byren JC, Caggana M, Carmichael SL, Cilliers D, Conway K, Crawford K, Cuellar A, Di Rocco F, Engel M, Fearon J, Feldkamp ML, Finnell R, Fisher S, Freudlsperger C, Garcia-Fructuoso G, Hagge R, Heuze Y, Harshbarger RJ, Hobbs C, Howley M, Jenkins MM, Johnson D, Justice CM, Kane A, Kay D, Gosain AK, Langlois P, Legal-Mallet L, Lin AE, Mills JL, Morton JEV, Noons P, Olshan A, Persing J, Phipps JM, Redett R, Reefhuis J, Rizk E, Samson TD, Shaw GM, Sicko R, Smith N, Staffenberg D, Stoler J, Sweeney E, Taub PJ, Timberlake AT, Topczewska J, Wall SA, Wilson AF, Wilson LC, Boyadjiev SA, Wilkie AOM, Richtsmeier JT, Jabs EW, Romitti PA, Karasik D, Birnbaum RY, Peter I. Regulatory elements in SEM1-DLX5-DLX6 (7q21.3) locus contribute to genetic control of coronal nonsyndromic craniosynostosis and bone density-related traits. Genet Med Open. 2024;2:101851. doi: 10.1016/j.gimo.2024.101851. Epub 2024 May 17. PMID 39345948
- [Result] Lesciotto KM, Motch Perrine SM, Kawasaki M, Stecko T, Ryan TM, Kawasaki K, Richtsmeier JT. Phosphotungstic acid-enhanced microCT: Optimized protocols for embryonic and early postnatal mice. Dev Dyn. 2020 Apr;249(4):573-585. doi: 10.1002/dvdy.136. Epub 2019 Nov 28. PMID 31736206
- [Result] Lee C, Richtsmeier JT, Kraft RH. A MULTISCALE COMPUTATIONAL MODEL FOR THE GROWTH OF THE CRANIAL VAULT IN CRANIOSYNOSTOSIS. Int Mech Eng Congress Expo. 2014 Nov;2014:V009T12A061. doi: 10.1115/IMECE2014-38728. PMID 25909093
- See also: The eMOSS staging system-free, public webtool for any PI requiring increased temporal resolution for research using embryonic mice. Developed thru a collaboration-Dr. Joan Richtsmeier lab, Penn State Univ & Dr. James Sharpe lab, Center for G — http://limbstaging.crg.es/